CLINICAL TRIAL: NCT03243539
Title: Implementation of Neuro Lung Protective Ventilation in Patients With Acute Brain Injury
Brief Title: Implementation of Neuro Lung Protective Ventilation
Acronym: NEUROVENT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colin Grissom (Other)
Responsible Party: Sponsor-Investigator, Colin Grissom, Co-Medical Director Shock Trauma ICU, Intermountain Health Care, Inc.
Organization: Intermountain Health Care, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1050582
Record Dates: First submitted 2017-07-14; First posted 2017-08-09 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Acute Brain Injury; Traumatic Brain Injury; Intracerebral Hemorrhage; Stroke; Cerebral Edema; Anoxic Brain Injury
Keywords: lung protective ventilation
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Cerebral Hemorrhage; Stroke; Brain Edema; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Protective Ventilation (Experimental): Subjects with acute brain injury (traumatic brain injury and non-traumatic brain injury) will receive neuro lung protective ventilation which targets a normal arterial partial pressure of carbon dioxide with the lowest tidal volume possible (6 to 8 ml/kg predicted body weight). Protocols for oxygenation and weaning from the ventilator will also be followed.
  Interventions: Procedure: Lung Protective Ventilation

INTERVENTIONS:
Procedure: Lung Protective Ventilation — Neuro lung protective ventilation for patients with acute brain injury is designed to target a normal partial pressure of arterial carbon dioxide and decrease initial tidal volumes toward a target 6 ml/kg predicted body weight PBW (range 6 to 8 ml/kg PBW)

SUMMARY:
Patients who experience lung injury are often placed on a ventilator to help them heal; however, if the ventilator volume settings are too high, it can cause additional lung injury. It is proven that using lower ventilator volume settings improves outcomes. In patients with acute brain injury, it is proven that maintaining a normal partial pressure of carbon dioxide in the arterial blood improves outcomes. Mechanical ventilator settings with higher volumes and higher breathing rates are sometimes required to maintain a normal partial pressure of carbon dioxide. These 2 goals of mechanical ventilation, using lower volumes to prevent additional lung injury but maintaining a normal partial pressure of carbon dioxide, are both important for patients with acute brain injury. The investigators have designed a computerized ventilator protocol in iCentra that matches the current standard of care for mechanical ventilation of patients with acute brain injury by targeting a normal partial pressure of carbon dioxide with the lowest ventilator volume required.

This is a quality improvement study with the purpose of observing and measuring the effects of implementation of a standard of care mechanical ventilation protocol for patients with acute brain injury in the iCentra electronic medical record system at Intermountain Medical Center. We hypothesize that implementation of a standardized neuro lung protective ventilation protocol will be feasible, will achieve a target normal partial pressure of carbon dioxide, will decrease tidal volumes toward the target 6 mL/kg predicted body weight, and will improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Acute brain injury due to non-traumatic causes (stroke, spontaneous intracranial hemorrhage, cerebral edema, anoxic brain injury) or traumatic brain injury.
2. Initiation of mechanical ventilation in the emergency department or intensive care unit at an Intermountain Healthcare hospital
3. Age ≥ 18 years

Exclusion Criteria:

1. Transition to comfort care in the emergency department or on the same day of admission to the ICU
2. Death on the same day of admission to the emergency department or ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Level Proportion of time on Mechanical Ventilation with a Tidal Volume <= 6.5 ml/kg PBW | Time of initiation of mechanical ventilation to time of cessation of mechanical ventilation, an average of 5 days

SECONDARY OUTCOMES:
Proportion of time with a target PaCO2 of 35 to 45 mm Hg | Time of initiation of mechanical ventilation to time of cessation of mechanical ventilation, an average of 5 days
Average number of protocol deviations for all subjects (protocol compliance) | Time of initiation of mechanical ventilation to time of cessation of mechanical ventilation, an average of 5 days
  Average of the number of instances in which the procedures specified in the protocol were not followed for each enrolled subject
Hospital Discharge Disposition | Day of hospital discharge, an average of 10 days after admission
  Routine, skilled nursing facility, home health, other
Hospital, 28-Day, and 90-Day Mortality | Hospital admission through 90 days
Ventilator-free days to day 28 | Initiation of mechanical ventilation to day 28
Time to First ICU Activity | Day of admission to day of first ICU activity, an average of 0.2 days
Hospital, ICU Length of Stay | Day of admission to day of discharge, an average of 10 days
Health Care Utilization | Day of admission to day of discharge, an average of 10 days
  Number of procedures/surgeries while in the hospital and number of days of hospitalization
Quality of Life - up to 1 year after day of discharge | Day of admission until up to 1 year after day of discharge
  May include SF-36 or similar measures
Costs of Care | Day of admission to day of discharge, an average of 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Colin K Grissom, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No
The intent of the investigators is to publish their experience with implementation of this protocol in the peer reviewed medical literature.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03243539/Prot_SAP_000.pdf